CLINICAL TRIAL: NCT06810986
Title: Phase 2 Research Study for Type 2 Diabetes Mellitus Through Digital Therapeutics
Brief Title: Cohort Study Evaluating Glycaemic Control in Individuals with Type 2 Diabetes Mellitus Through Digital Therapeutics (DM DTx)
Acronym: DM DTx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EVYD Technology (Industry)
Collaborators: Ministry of Health, Brunei Darussalam (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MHREC/MOH/2024/11; BALANCE Programme (Other: EVYD Technology)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Lifestyle Intervention; Digital Therapeutics; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital Therapeutics for Type 2 Diabetes Mellitus (Experimental): 16 weeks digital intervention with online support
  This study is a single-arm, non-randomised clinical trial, which will collect participant's baseline data, apply relevant assessment scales, collect data using a comprehensive digital intervention in 16 weeks to evaluate the improvement of relevant markers post intervention.
  Interventions: Behavioral: 16-week digital intervention

INTERVENTIONS:
Behavioral: 16-week digital intervention — Participants will be enrolled in a 16-week programme with the aim to manage T2DM through lifestyle adjustments. Participants will be given online support by their personal health coach with additional support from a dietitian or clinician in the study if required.
  Each participant will receive personalised recommendations for blood glucose monitoring schedule, diet and physical activity. Participants are required to log their blood glucose, diet and physical activity in the BruHealth application. Participants will review their progress with their health coach via video consultation on a regular basis. Additionally, participants will also participate in a structured diabetes self-management education course.
  Other Names: Lifestyle Intervention

SUMMARY:
This study is conducted to evaluate the effectiveness of Digital therapeutics (DTx) in managing patients with Type 2 Diabetes Mellitus (T2DM) by delivering digital lifestyle interventions through a national health application (BruHealth).

DETAILED DESCRIPTION:
This study is a single-arm, non-randomised clinical trial designed to evaluate the effectiveness and feasibility of an online management approach to improve glycaemic control in individuals with Type 2 Diabetes Mellitus (T2DM) through a digital lifestyle intervention (named the BALANCE Programme) over a 16-week period. The intervention leverages the Diabetes Mellitus Digital Therapeutics (DM DTx) module within the BruHealth application. Additionally, a Healthcare Professional (HCP) portal is included to facilitate ongoing monitoring and support, ensuring personalized care and real-time interactions between participants and healthcare providers.

In addition, Muslim participants are offered the option of providing information in the DM DTx module about their fasting practices during Ramadan as an opportunistic way of obtaining data on the fasting risk and fasting experience in this cohort.

Primary Objective:

The primary objective is to assess the proportion of participants who experience a reduction in HbA1c levels by at least 0.6% by the end of the 16-week intervention period.

Secondary Objectives:

1. To evaluate the overall changes in HbA1c, fasting blood glucose, Body Mass Index (BMI), waist circumference and improvements in lipid profile components (such as cholesterol and triglycerides) at week 16, compared to baseline measurements;
2. To evaluate participants' feedback on their experience with the BALANCE Programme and its usability after 16 weeks of usage;
3. to evaluate fasting experience amongst Muslims with T2DM during Ramadhan and to calculate their fasting risk using IDF-DAR score.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Diagnosed with T2DM who are on any one or more of the following treatments:

  1. oral glucose lowering medication(s)
  2. any type of insulin treatment (up to 2 injections a day only)
  3. on diet control only
  4. GLP-1 receptor agonist established at least 6 months prior to enrolment

Exclusion Criteria:

* Diagnosed with T2DM on more than 2 insulin injections a day
* Diagnosed with Type 1 Diabetes Mellitus (T1DM)
* Pregnant / Breast-feeding
* Recent Myocardial Infarction (MI) or Stroke / Cerebrovascular Accidents (CVA) in the past 6 months
* Heart failure
* Liver failure
* Active cancer
* Undergoing active treatment for active foot disease
* Undergoing active treatment for active diabetes-related eye disease
* CKD stage 4 and 5 (eGFR < 30ml/min)
* Hospitalisation for any reason in the past 6 months
* Advised by doctor to not participate in intense physical activity
* Physical disability and/or unable to perform Activities of Daily Living (ADL) independently
* Unable to use Youtube on mobile devices
* Unable to use BruHealth independently

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in HbA1c from baseline following a 16-week lifestyle intervention | 16 weeks
  The proportion of participants who achieve at least 0.6% reduction in HbA1c from baseline following a 16-week lifestyle intervention provided by DM DTx

SECONDARY OUTCOMES:
Overall change in HbA1c | 16 weeks
  Evaluation of overall changes in HbA1c
Change in fasting lipid profile | 16 weeks
  Evaluation of overall changes in fasting lipid profile
Change in fasting blood glucose | 16 weeks
  Evaluation of overall changes in fasting blood glucose
Change in BMI | 16 weeks
  Evaluation of overall changes in BMI
Change in waist circumference | 16 weeks
  Evaluation of overall changes in waist circumference
Participants' feedback on the use of DM DTx | 16 weeks
  Evaluation of participants' feedback of DM DTx through a series of questionnaires completed on end line

CONTACTS AND LOCATIONS:
Overall Officials: Chong Pui Lin, BM, MD, Principal Investigator — Raja Isteri Pengiran Anak Saleha (RIPAS) hospital
Locations (1):
- EVYD Technology, Bandar Seri Begawan, Brunei